CLINICAL TRIAL: NCT05532878
Title: Pharmacokinetics and Safety Profile of Apixaban in Patients With Peritoneal Dialysis
Brief Title: Pharmacokinetics of Apixaban in Peritoneal Dialysis
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Department of Medicine & Therapeutics, Chinese University of Hong Kong
Other Study IDs: CRE-2020.284
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation
Keywords: peritoneal dialysis
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: stable PD patients with non-valvular AF
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Apixaban 2.5 mg daily

SUMMARY:
Atrial fibrillation (AF) is fairly prevalent in patients with end stage renal disease (ESRD) with the prevalence estimated to be 3.8 - 27%. While it is reported that patient with peritoneal dialysis (PD) has a lower incidence of AF as compared to patient with haemodialysis (HD), the risk is still substantially higher than in the general population. AF is a known risk factor for embolic stroke and stroke causes significant morbidity and mortality. Anticoagulation in an effective treatment for the prevention of stroke in the general population. However, this is less clear in the ESRD populations.

Despite the risk of stroke is higher than general population, the management of AF in patients with ESRD remains controversial with limited and often conflicting result for the use of traditional vitamin K antagonists. It also showed an increased risk of bleeding with the use in ESRD patients.

With the advent of direct oral anticoagulants (DOACs), there is growing interest in advocating their uses and studies have been done to assess their safety profile. In fact, several randomized control trials are being performed. However, these studies are done in HD populations and there is no data for PD populations at all so far.

Given the physiology of drug clearance is different between the two renal replacement modalities, the investigators purpose to assess the pharmacokinetics and the safety profile of Apixaban in PD populations. By establishing the pharmacokinetics and its safety profile, apixaban may be a more attractive option for anticoagulation for AF or other venous thrombotic indications in PD population.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is fairly prevalent in patients with end stage renal disease (ESRD) with the prevalence estimated to be 3.8 - 27%. While it is reported that patient with peritoneal dialysis (PD) has a lower incidence of AF as compared to patient with haemodialysis (HD), the risk is still substantially higher than in the general population. AF is a known risk factor for embolic stroke and stroke causes significant morbidity and mortality. Anticoagulation in an effective treatment for the prevention of stroke in the general population. However, this is less clear in the ESRD populations.

Despite the risk of stroke is higher than general population, the management of AF in patients with ESRD remains controversial with limited and often conflicting result for the use of traditional vitamin K antagonists. It also showed an increased risk of bleeding with the use in ESRD patients.

With the advent of direct oral anticoagulants (DOACs), there is growing interest in advocating their uses and studies have been done to assess their safety profile. In fact, several randomized control trials are being performed. However, these studies are done in HD populations and there is no data for PD populations at all so far.

Given the physiology of drug clearance is different between the two renal replacement modalities, the investigators purpose to assess the pharmacokinetics and the safety profile of Apixaban in PD populations. By establishing the pharmacokinetics and its safety profile, apixaban may be a more attractive option for anticoagulation for AF or other venous thrombotic indications in PD population.

ELIGIBILITY:
Inclusion Criteria:

* stable PD patients with non-valvular AF and with no significant residual renal function

Exclusion Criteria:

* increased risk of bleeding and those with contraindications to anticoagulation such as history of gastrointestinal bleeding, dual anti-platelet therapy, active malignancy, recent trauma and stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stable PD patients with non-valvular AF and with no significant residual renal function
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Apixabn level | 0 to 12 hours (14 time points)
  Blood anti-factor Xa activity

CONTACTS AND LOCATIONS:
Overall Officials: Winston WS Fung, MBBS, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No personal data will be shared.